CLINICAL TRIAL: NCT03007693
Title: A Randomized, Placebo-controlled, Double-blind, Multiple Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ 61393215 in Healthy Subjects
Brief Title: A Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ 61393215 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: CR108250; 2016-003894-16 (EudraCT Number); 61393215EDI1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-12-30; First posted 2017-01-02 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JNJ-61393215 (Multiple Ascending Dose Phase) (Experimental): Participants will receive JNJ- 61393215 once daily for 7 days. 4 sequential cohorts will be enrolled to evaluate escalating doses which will be defined, based on safety, tolerability and pharmacokinetic (PK) data from the preceding cohorts. Dose adjustment/selection (increase/decrease) for the next cohort will be based on the JNJ- 61393215 PK profile up to and including the last day of dosing (24 hours postdose) and the safety and tolerability profile of the current cohort.
  Interventions: Drug: JNJ-61393215
- Placebo (Multiple Ascending Dose Phase) (Placebo Comparator): Participants will receive JNJ- 61393215 matching placebo for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-61393215 — Participants will receive JNJ-61393215 for 7 days.
  Arms: JNJ-61393215 (Multiple Ascending Dose Phase)
Drug: Placebo — Participants will receive JNJ- 61393215 matching placebo for 7 days.
  Arms: Placebo (Multiple Ascending Dose Phase)

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of JNJ-61393215 after multiple consecutive dose administrations and to characterize the pharmacokinetics (PK) of JNJ-61393215 in plasma after multiple consecutive dose administrations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants between 18 and 55 years of age, inclusive
* Participants must have a body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2), inclusive (BMI = weight/height square)
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead ECG [incl. QTcF less than or equal to [<=] 450 milliseconds (msec) for males] performed at screening and admission to the clinical unit. Minor abnormalities in electrocardiogram (ECG), which are not considered to be of clinical significance by the investigator, are acceptable. The presence of Left Bundle Branch Block (LBBB), AV Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator [ICD] will lead to exclusion
* Participants must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the Participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the Participant's source documents and initialed by the investigator
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of contraception e.g., either condom with spermicidal foam/gel/film/cream/suppository during the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug. All men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partner should also use a highly effective method of contraception for at least the same duration. Examples of highly effective contraceptives include implantable progestogen-only hormone contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); vasectomized partner; sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.), combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, and transdermal; progestogen-only hormone contraception associated with inhibition of ovulation: oral and injectable.
* Participants must be willing to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Participant has a history of or current liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness, though minor deviations, which are not considered to be of clinical significance to both the investigator and to the Janssen Safety Responsible Physician, are acceptable
* Current or past history of any psychiatric disorder as classified according to Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) or DSM-V, with the exclusion of an anxiety disorder (i.e., panic disorder with or without agoraphobia, social anxiety disorder, and generalized anxiety disorder)
* Participant has any liver function test (including alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyltransferase [gGT], alkaline phosphatase [ALP and bilirubin] at screening exceeding the upper limit of normal
* Participant has estimated glomerular filtration rate (eGFR) <60 milliliter per minute (mL/min)/1.73m^2 at screening (provided by the local laboratory)
* Participant has a heart rate < 50 beats per minute (bpm) or > 100 bpm or systolic blood pressure greater than or equal to (>=) 150 millimeter of mercury (mmHg) at screening or at admission to the clinical unit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events as a Measure of Safety and Tolerability | up to 4 weeks
Time To Reach The Maximum Plasma Concentration (Tmax) | Day 1
  Tmax is time to reach the maximum plasma concentration.
Maximum Plasma Concentration (Cmax) | Day 1
  Cmax is maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time [0 to24] (AUC[0-24]) | Day 1
  AUC[0-24] is area under the plasma concentration- time curve from time [0 to 24].
The Observed Plasma Concentration Just Prior To the Beginning or at the End of a Dosing Interval of any Dose Other Than the First Dose (Ctrough) | Days 2 to 6
  Ctrough is the observed plasma concentration just prior to the beginning or at the end of a dosing interval of any dose other than the first dose.
The Observed Plasma Concentration Just Prior To the Beginning or at the End of a Dosing Interval of any Dose Other Than the First Dose (Ctrough) | Day 7
  Ctrough is the observed plasma concentration just prior to the beginning or at the end of a dosing interval of any dose other than the first dose.
Minimum Observed Plasma Concentration During Dosing Interval (tau) (Cmin) | Day 7
  Cmin is minimum observed plasma concentration during dosing interval (tau).
Time To Reach The Maximum Plasma Concentration (Tmax) | Day 7
  Tmax is time to reach the maximum plasma concentration.
Maximum Plasma Concentration (Cmax) | Day 7
  Cmax is maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time [0 to24] (AUC[0-24]) | Day 7
  AUC[0-24] is Area under the plasma concentration- time curve from time [0 to 24].
Average Plasma Concentration at Steady State Over the Dosing Interval (Cavg) | Day 7
  Cavg is average plasma concentration at steady state over the dosing interval.
Fluctuation Index (FI) | Day 7
  Fluctuation Index is defined as percentage of fluctuation, calculated as: 100*([Cmax-Cmin]/Cavg).
Total Apparent Oral Clearance, Calculated as Dose/AUCtau at Steady-State (CL/F) | Day 7
  CL/F is total apparent oral clearance, calculated as dose/AUCtau at steady-state.
Apparent Terminal Elimination Rate Constant, Determined By Linear Regression of the Terminal Points of the Ln-Linear Plasma Concentration-Time Curve (Lambda[Z]) | Day 7
  Lambda[Z] is apparent terminal elimination rate constant, determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Apparent Elimination Half-Life Associated With The Terminal Slope of The Semilogarithmic Drug Concentration-Time Curve, After Multiple-Dose Administration Only (t1/2term) | Day 7
  T1/2term is apparent elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve, after multiple-dose administration only.
Ratio of Maximum Plasma Concentration (Cmax) Test (Day 7 [steady-state]/ref (Day 1) (Ratio Cmax,test/ref) | Day 7
  Ratio Cmax,test/ref is ratio of maximum plasma concentration (Cmax) test (day 7 [steady-state]/ref (day 1).
Ratio of Area Under the Plasma Concentration-Time Curve From Time [0 to24] (AUC[0-24]) Test (Day 7 [steady-state]/ref (Day 1) (Ratio AUC24h,test/ref) | Day 7
  Ratio AUC24h,test/ref is ratio of area under the plasma concentration- time curve from time [0 to 24] (AUC[0-24]) test (day 7 [steady-state]/ref (day 1).

SECONDARY OUTCOMES:
Effect of JNJ-61393215 on Alertness/Sedation Through the Bond & Lader Visual Analogue Scale | Day 1 and Day 7
  Visual Analogue Scale (VAS) is made up of 16 pairs of alternative descriptors of mood and attention at either end. The Bond-Lader of a 10 cm line. Participants will rate their feelings at the time of assessment by indicating the point on the line which best represent their mood. Each item is scored by measuring the position relative to the left hand end of the line and levels of anxiety, sedation, and dysphoria are then calculated from the combined scores of selected items. The score ranges from 0 to 100, with a high score reflecting a high level of anxiety, sedation or dysphoria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Leiden, Netherlands